CLINICAL TRIAL: NCT05929274
Title: Safety and Efficacy of Transcranial Direct Current Stimulation in Pediatric Disorders of Consciousness
Brief Title: Safety and Efficacy of tDCS in Pediatric DoC
Acronym: tDCS-DoC-Ped
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has never started because of internal decisions
Sponsor: Giovanna Cristella (Other)
Responsible Party: Sponsor-Investigator, Giovanna Cristella, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Organization: Fondazione Don Carlo Gnocchi Onlus (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS-DoC-Ped
Record Dates: First submitted 2023-05-09; First posted 2023-07-03 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Disorder of Consciousness
Keywords: Pediatric population; tDCS; disorder of consciousness
MeSH Terms: conditions — Consciousness Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Using a sham-controlled randomized double-blind design, 10 patients were randomly assigned to group A or B.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Comparator - real tDCS (Experimental): real tDCS: anodal transcranial direct current stimulation were delivered over the left DLPF cortex in patients
  Interventions: Device: tDCS
- Sham Comparator - sham tDCS (Sham Comparator): sham transcranial direct current stimulation were delivered over the left DLPF cortex in patients.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — Direct current was applied by a battery-driven constant current stimulator using saline-soaked surface sponge electrodes (7 3 5 cm) with the anode positioned over the left dorsolateral prefrontal cortex (F3 according to the 10-20 international system for EEG placement) and the cathode placed over the right supraorbital region. During real tDCS, the current was increased to 2 milliampere (mA) from the onset of stimulation and applied for 20 minutes.
  Arms: Active Comparator - real tDCS
Device: sham tDCS — For the sham condition (sham tDCS), the same electrode placement was used as in the stimulation condition, but the current was applied for only 5 seconds, and was then ramped down.
  Arms: Sham Comparator - sham tDCS

SUMMARY:
Background: Despite established evidence supporting the use of tDCS in the adult patient with disorders of consciousness, its use in paediatric patients with brain injury is still limited. Regarding the use of tDCS in paediatric patients with DoC, the scientific evidence still appears to be preliminary about the safety profile and requires further data before investigating efficacy on a broad scale. In fact, although the method has been shown to be safe in other clinical conditions, efficacy and tolerability in children with DoC may vary significantly depending on differences in activation threshold and the presence of underlying pathological electrical activity The implementation of clinical trials investigating the safety and tolerability of tDCS in paediatric patients with DoC now represents an essential first step for a future determination of the efficacy of this method in a population for which therapeutic options are currently extremely limited Objective: The study aim to verify the safety of tDCS treatment and to evaluate the effectiveness of stimulation of the left dorsolateral prefrontal cortex by tDCS in promoting improvement in the level of consciousness in paediatric patients with Disorders of Consciousness.

Method: in this mono-center, randomised, double blind cross-over controlled pilot study, real or sham tDCS were applied to the left dorsolateral prefrontal (DLPF) cortex of paediatric patients with disorders of consciousness for two weeks, followed by two weeks of washout, then real or sham tDCS were applied to the left dorsolateral prefrontal (DLPF) cortex for other two weeks, followed by another two weeks of washout.

DETAILED DESCRIPTION:
Introduction Following a severe acquired brain injury of traumatic, hypoxic-anoxic, or vascular origin, conditions of very severe cognitive and motor impairment can occur, named as Disorders of Consciousness (DoC), which include the Vegetative State (VS), characterized by the presence of vegetative functions 'in absence of self-awareness and awareness of the environment, and the Minimal Consciousness State (MCS), in which minimal, inconstant, but repeated behavioral responses to visual, verbal or nociceptive stimuli are recognizable, clearly distinguishable from reflex responses.

Differential diagnosis can be complex, and one of the first (and most frequent) sign of transition from VS to MCS is the appearance of visual tracking of salient stimuli .The natural evolution of DoC is influenced by the etiology, being anoxic forms less favorable to recover than other forms. It has been proven that patients with MCS have more favorable prognoses than patients with VS, especially when the condition of MCS occurs within a few months from the acute event.

Despite significant improvement in the understanding of the neural correlates of DoC, the treatment options currently available for these patients are still very limited. Recent findings, however, suggest a broad spectrum of therapeutic possibilities. In the last decade, in fact, several studies have reported signs of spontaneous improvement of consciousness a few years after the acute event in some patients diagnosed with VS .Furthermore, studies on treatments that enhance cognitive abilities in patients with DoC have shown that deep brain stimulation (DBS) in the intralaminar nuclei of the thalamus and some drugs such as amantadine , intrathecal baclofen and zolpidem can improve sign of consciousness behavior in a large cohort of acute and sub-acute patients with DoC of traumatic origin in sham-controlled studies.

In pediatric population with DoC, the exact incidence of VS and MCS is not entirely clear; however, it appears that MCS is more frequent condition than VS compared to adult patients After the acute phase, the pediatric DoC patient starts a specific rehabilitation pathway; its primary goal is the maximum possible recovery of consciousness. During intensive rehabilitation, about 2/3 of pediatric and young adult patients emerges to a state of consciousness within 7 months after the acute event. The rehabilitation program includes a neuropsychological approach dedicated to the recovery of consciousness; from a pharmacological point of view, the literature suggests the use of the following drugs for pediatric DoC: carbidopa-levodopa, amantadine, zolpidem, and methylphenidate.

Efficacy During the last 20 years, intervention studies with innovative non-invasive brain stimulation techniques, such as transcranial direct current stimulation (tDCS), have shown that cycles of low-intensity electrical stimulation delivered via electrodes applied to the scalp in specific areas can promote the processes of neuronal plasticity, i.e. the ability of the central nervous system to modify its structure and functioning in response to new information and experiences. These effects appear to be particularly interesting in the treatment of various neurological and psychiatric disorders such as Parkinson's Disease, post-stroke aphasia or the neuropsychological outcomes of Multiple Sclerosis. More recently, tDCS has been shown to be a safe, inexpensive, and simple technique that can be easily integrated into rehabilitation programs. In particular, stimulation with tDCS has been shown to be effective in aiding the recovery of the state of consciousness in the adult population in the acute, subacute and chronic phase, predominantly in the MCS condition, considering traumatic and non-traumatic etiology. This occurs especially in the anodic stimulation mode of the left dorsolateral prefrontal cortex. In a study in which tDCS was applied for five consecutive days on the motor cortex and left prefrontal cortex in 10 chronic DoC patients, the effect of stimulation was evaluated up to 12 months after its ending, showing that even chronic DoC patients show signs of improvement and that this effect can be maintained up to 12 months after tDCS treatment. From a neurophysiological point of view, tDCS acts by increasing neuronal excitability and facilitating the action potential by modifying the excitability of N-methyl-D-aspartate (NMDA) receptors. In addition, tDCS can enhance active synaptic connections. The effect of a single tDCS session lasts approximately 60 to 90 minutes; when stimulation is repeated 10 times up to 20 sessions it has been found that the effects last up to 3 months after the ending of the stimulation sessions.

Security The safety and tolerability of tDCS have been widely demonstrated in adult patients with consciousness disorders and brain damage. Most authors have found a very good safety profile in patients with DoC, recording adverse effects that are generally transient and mild. Common adverse effects reported during or immediately after tDCS include tingling or numbness in stimulated skin, headache, nausea and fatigue. In addition, there is currently no evidence of long-term adverse or serious adverse effects associated with the use of tDCS in adult DoC patients.

The possibility of subclinical neuronal damage induced by stimulation has been ruled out in studies that assessed serum levels of neuron-specific enolase (NSE, a marker of neuronal damage) before and after stimulation and by studies with EEG or magnetic resonance imaging. Regarding the protocols utilized, this method has to be regarded as safe.

Despite established evidence supporting the use of tDCS in the adult patient, its use in paediatric patients with brain injury is still limited. To date, tDCS is mainly used in paediatric age as a complementary therapy in the rehabilitation of neurodevelopmental disorders such as infantile cerebral palsy, attention deficit hyperactivity disorder (ADHD), obsessive-compulsive disorder. In these patients, tDCS was confirmed to be a safe and well-tolerated technique even in the paediatric population with a small number of reported mild and short-lasting adverse events such as tingling (18%), discomfort (8%) and itching (7%).

Regarding the use of tDCS in paediatric patients with DoC, the scientific evidence still appears to be preliminary about the safety profile and requires further data before investigating efficacy on a broad scale. In fact, although the method has been shown to be safe in other clinical conditions, efficacy and tolerability in children with DoC may vary significantly depending on differences in activation threshold and the presence of underlying pathological electrical activity. The implementation of clinical trials investigating the safety and tolerability of tDCS in paediatric patients with DoC now represents an essential first step for a future determination of the efficacy of this method in a population for which therapeutic options are currently extremely limited. Lastly, several studies have shown that certain quantitative measures of functional connectivity derived from electroencephalographic and evoked-potential analysis (e.g., coherence of the EEG signal, presence of event-related evoked potentials) are capable of faithfully reflecting changes in the state of consciousness in adult DoC patients, contributing to the formulation of prognosis and the identification of patients who are most likely to benefit from treatment. In this sense, the identification of possible paediatric neurophysiological biomarker can help to provide a preliminary quantitative measure of response to treatment, while contributing to the understanding of the effect of tDCS on involved brain networks.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 4 and 17;
* prolonged condition (>3 and <12 months) of MCS and VS by severe brain injury;
* admission to the paediatric rehabilitation department of the Don Carlo Gnocchi Foundation in Florence;
* central nervous system drug therapy stable for at least one week;
* stable DoC (i.e. no change in DoC diagnosis detected by 2 consecutive CRS-Rs performed one week apart);
* Signature of informed consent by the legal representative.

Exclusion Criteria:

* Presence of extensive focal lesions in the left dorsolateral prefrontal cortex (DLPFC);
* radiological evidence of blood collection/liquid collection/other between the DLPFC and the anode placement site;
* seizures in the previous month;
* seizures and/or intermittent epileptiform discharges observed at the extended EEG during the screening phase or at any of the EEG recordings during participation in the study;
* Presence of established pregnancy;
* History of cranial surgery, presence of metallic, cochlear or electronic brain implant in the head or neck area, or ventricular shunt to pacemaker;
* Need for mechanical daytime ventilation;
* Head circumference less than 43 cm;
* bilateral severe or profound hypoacusia;
* Presence of skin lesions in the area to be stimulated;
* Taking sedative drugs and/or Na or Ca channel blockers or NMDA receptor antagonists presence of peritoneal ventricle shunt in the stimulated area (prefrontal cortex);
* serious clinical conditions that may influence the clinical diagnosis (e.g. severe liver failure or kidney).

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Evaluating the safety of tDCS treatment assessing the change over time | baseline (1-7 days), post-stimulation (within 30-minutes), follow-up (24 hours, 48 hours, 5 days)
  the ratio of reported adverse events between the two treatment groups and the proportion of treatments discontinued for adverse events will be assessed, using an "Adverse Event Collection Form" completed by a practitioner other than the parents will be used
Assessing the change of tolerability of treatment with tDCS | Baseline (1-7 days), pre-during-post stimulation (pre-stimulation: within 30 minutes, during: within 20 minutes, post-stimulation: within 30-minutes)
  Face, Legs, Activity, Cry and Consolability Scale (FLACC 0-10 worst value) scale will be used to assess tolerability of treatment
Assessing the change in the state of consciousness by using tDCS | days 1, 8, 12, 19, 35, 40, 47, 62, 92
  Coma Recovery Scale - Revised (CRS-R 0-23 best value) will be used to evaluate the effectiveness of tDCS

SECONDARY OUTCOMES:
To evaluate the effect of tDCS stimulation on brain electrical activity | days 1, 8, 35, 47, 62, 92
  analysis of EEG signal coherence measurements before and after the stimulation cycle
To evaluate the effect of tDCS stimulation on cortical electrical activity | days 1, 8, 35, 47, 62, 92
  cortical components analysis of event-related potentials (ERPs) before and after the stimulation cycle;
To evaluate the effect of tDCS stimulation in determining haemodynamic response (HDR) changes quantifiable | days 8, 35, 47, 62, 92
  Functional Near Infrared Spectroscopy (fNlRS): spectroscopic analysis at the level of stimulated areas after treatment
Assess caregiver satisfaction with the treatment | days 19 and 47
  Family Feedback Form Questionnaire will be submitted to caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Cristella, MD, Principal Investigator — IRCCS Fondazione Don Carlo Gnocchi ONLUS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung MG, Lo WD. Noninvasive brain stimulation: the potential for use in the rehabilitation of pediatric acquired brain injury. Arch Phys Med Rehabil. 2015 Apr;96(4 Suppl):S129-37. doi: 10.1016/j.apmr.2014.10.013. Epub 2014 Nov 6. PMID 25448248
- [Background] Elbanna ST, Elshennawy S, Ayad MN. Noninvasive Brain Stimulation for Rehabilitation of Pediatric Motor Disorders Following Brain Injury: Systematic Review of Randomized Controlled Trials. Arch Phys Med Rehabil. 2019 Oct;100(10):1945-1963. doi: 10.1016/j.apmr.2019.04.009. Epub 2019 May 10. PMID 31078616
- [Background] Estraneo A, Pascarella A, Moretta P, Masotta O, Fiorenza S, Chirico G, Crispino E, Loreto V, Trojano L. Repeated transcranial direct current stimulation in prolonged disorders of consciousness: A double-blind cross-over study. J Neurol Sci. 2017 Apr 15;375:464-470. doi: 10.1016/j.jns.2017.02.036. Epub 2017 Feb 17. PMID 28320187
- [Background] Giacino JT, Whyte J, Bagiella E, Kalmar K, Childs N, Khademi A, Eifert B, Long D, Katz DI, Cho S, Yablon SA, Luther M, Hammond FM, Nordenbo A, Novak P, Mercer W, Maurer-Karattup P, Sherer M. Placebo-controlled trial of amantadine for severe traumatic brain injury. N Engl J Med. 2012 Mar 1;366(9):819-26. doi: 10.1056/NEJMoa1102609. PMID 22375973
- [Background] Hameed MQ, Dhamne SC, Gersner R, Kaye HL, Oberman LM, Pascual-Leone A, Rotenberg A. Transcranial Magnetic and Direct Current Stimulation in Children. Curr Neurol Neurosci Rep. 2017 Feb;17(2):11. doi: 10.1007/s11910-017-0719-0. PMID 28229395
- [Background] Palm U, Segmiller FM, Epple AN, Freisleder FJ, Koutsouleris N, Schulte-Korne G, Padberg F. Transcranial direct current stimulation in children and adolescents: a comprehensive review. J Neural Transm (Vienna). 2016 Oct;123(10):1219-34. doi: 10.1007/s00702-016-1572-z. Epub 2016 May 12. PMID 27173384
- [Background] Saleem GT, Ewen JB, Crasta JE, Slomine BS, Cantarero GL, Suskauer SJ. Single-arm, open-label, dose escalation phase I study to evaluate the safety and feasibility of transcranial direct current stimulation with electroencephalography biomarkers in paediatric disorders of consciousness: a study protocol. BMJ Open. 2019 Aug 10;9(8):e029967. doi: 10.1136/bmjopen-2019-029967. PMID 31401607